CLINICAL TRIAL: NCT01127178
Title: Phase 1 Study of the Poly (ADP-Ribose) Polymerase Inhibitor E7016 in Combination With Temozolomide in Subjects With Advanced Solid Tumors
Brief Title: Study of Poly (ADP-Ribose) Polymerase (PARP) Inhibitor E7016 in Combination With Temozolomide in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic decision, which is unrelated to safety
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7016-A001-101
Record Dates: First submitted 2010-05-10; First posted 2010-05-20 (Estimated); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2015-12

CONDITIONS: Solid Tumors
MeSH Terms: interventions — 10-((4-hydroxypiperidin-1-yl)methyl)chromeno(4,3,2-de)phthalazin-3(2H)-one; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E7016 + TMZ (Experimental)
  Interventions: Drug: E7016 + TMZ

INTERVENTIONS:
Drug: E7016 + TMZ — Single-Dose PK Period (single oral dose of E7016 on Day -7) in the Dose-Escalation Component; Multiple-Dose Treatment Cycles (7 days of oral E7016 + 5 days of oral TMZ) added in Cycle 1 of the Dose-Escalation Component and in Cycles 1 through 6 of the Expansion Component.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of poly (ADP-Ribose) polymerase inhibitor E7016 when used with temozolomide (TMZ) in patients with advanced solid tumors and gliomas.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria may be included in the study.

1. Histopathologically confirmed melanoma or other solid tumors (excluding malignant brain tumors) for which no standard therapy is available (Dose-Escalation Component only). During the Expansion Component, enrollment will be restricted to subjects with histopathologically proven gliomas and will include subjects eligible for TMZ therapy as well as those who have failed TMZ therapy; and those who are either not appropriate candidates for radiation therapy or who refuse radiation therapy. Subjects who are taking either strong cytochrome P450 (CYP) inhibitors or inducers may be enrolled.
2. Life expectancy greater than or equal to 3 months after starting E7016.
3. Performance status (PS) 1 to 2 on the Eastern Cooperative Oncology Group (ECOG) scale.
4. Adequate renal function indicated by serum creatinine less than 1.5 mg/dL or calculated creatinine clearance greater than 50 mL/minute.
5. Adequate bone marrow reserve:

   1. ANC greater than or equal to 1500/mm3,
   2. Platelets greater than or equal to 100,000/mm3 (without transfusion),
   3. Hemoglobin greater than or equal to 10 g/dL (less than 10.0 g/dL is acceptable if corrected by growth factor or transfusion).
6. Adequate liver function:

   1. Bilirubin less than or equal to 1.5x the upper limit of normal (ULN) (less than or equal to 3 x ULN if subject has liver metastases),
   2. Alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 times ULN (less than or equal to 5 x ULN if subject has liver metastases).
7. Males and females age greater than or equal to 18 years at the time of informed consent.

   1. Female subjects of childbearing potential must have a negative serum beta human chorionic gonadotropin (BhCG) test at Visit 1 (Screening) and a negative urine pregnancy test prior to the first dose of E7016 capsules in the Single-Dose PK Period and again prior to the first dose of E7016 in Cycle 1.
   2. Male subjects who are partners of women of childbearing potential must use or their partners must use a highly effective method of contraception (eg, condom + spermicide, condom + diaphragm with spermicide, IUD) beginning at least 1 menstrual cycle prior to starting study drug(s), throughout the entire study period, and for 30 days after the last dose of study drug.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participation in the study:

1. Subjects with primary or metastatic brain tumors are excluded from the Dose-Escalation Component.
2. Subjects with active malignancies other than gliomas are excluded from the Expansion Component.
3. Subjects taking medications which are either strong CYP inhibitors or inducers will be excluded from the Dose-Escalation Component.
4. Prior treatment with a PARP inhibitor.
5. Inability to tolerate 150 mg/m2/d TMZ during previous therapy with TMZ.
6. Known allergy, hypersensitivity, or other contraindication to E7016, TMZ, or dacarbazine or any of the other components of the formulations.
7. Known human immunodeficiency virus infection, active hepatitis B or C.
8. Active infections requiring specific anti-infective therapy
9. Subjects who have had a major surgical procedure (including tumor resection) within 4 weeks prior to initiating E7016 treatment.
10. Subjects scheduled for surgery during the projected course of the study.
11. Females who are pregnant (positive B-hCG test) or breastfeeding.
12. Chemotherapy, radiation therapy, or immunotherapy within 4 weeks prior to initiating E7016 treatment (6 weeks for mitomycin C or nitrosoureas).
13. Prolongation of QTc interval (500 msec).
14. Achlorhydria or use of antacids, proton-pump inhibitors, or other drugs known to raise gastric pH within 2 weeks prior to study drug administration.
15. Any history of or concomitant medical condition or clinically significant disease making the subject medically unfit to receive the study drug or, in the opinion of the investigator, unsuitable for any other reason.
16. Unable to swallow multiple capsules.
17. History of drug or alcohol dependency or abuse within approximately the last 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03-29 (Actual); Primary Completion 2011-02-24 (Actual); Study Completion 2011-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Medical Services, Study Director — Eisai Medical Services
Locations (5):
- United States (5):
  - Boston, Massachusetts
  - Lebanon, New Hampshire
  - Greenville, South Carolina
  - San Antonio, Texas
  - Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 29 March 2010 to 24 February 2011.
Pre-assignment Details: A total of 13 participants were screened, of which 1 was screen failure and 12 were enrolled to receive study treatment in Dose Escalation Part. The study was terminated due to sponsor's strategic decision, which is unrelated to safety, therefore no participants were enrolled in the Dose Expansion part. Hence, no data collection and analysis were done during Dose Expansion part of this study.
Groups:
- Dose Escalation Part: E7016 4 mg/kg/Day + Temozolomide 150 mg/m^2: Participants received single oral dose of 4 milligrams per kilogram per day (mg/kg/day) E7016 capsule on Day -7 for pharmacokinetic (PK) analysis, followed by once daily dose from days 1 to 5 in combination with temozolomide 150 milligrams per square meter (mg/m^2) capsule and alone on days 6 and 7 of Cycle 1 (cycle length=28 days) in Treatment Phase. Participants who completed the Treatment Phase entered the Extension Phase of Dose Escalation Part and continued the treatment in Extension Phase in same manner of Treatment Phase until unacceptable toxicity, disease progression, termination by the treating investigator, withdrawal of consent, termination of the program by the sponsor, or treatment delay greater than (>) 2 weeks for recovery of toxicity.
- Dose Escalation Part: E7016 8 mg/kg/Day + Temozolomide 150 mg/m^2: Participants received single oral dose of 8 mg/kg/day E7016 capsule on Day -7 for PK analysis, followed by once daily dose from days 1 to 5 in combination with temozolomide 150 mg/m^2 capsule and alone on days 6 and 7 of Cycle 1 (cycle length=28 days) in Treatment Phase. Participants who completed the Treatment Phase entered the Extension Phase of Dose Escalation Part and continued the treatment in Extension Phase in same manner of Treatment Phase until unacceptable toxicity, disease progression, termination by the treating investigator, withdrawal of consent, termination of the program by the sponsor, or treatment delay >2 weeks for recovery of toxicity.
Period: Dose Escalation: Treatment Phase
Arm/Group | Dose Escalation Part: E7016 4 mg/kg/Day + Temozolomide 150 mg/m^2 | Dose Escalation Part: E7016 8 mg/kg/Day + Temozolomide 150 mg/m^2
Started | 9 | 3
Completed | 5 | 3
Not Completed | 4 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 2 | 0
Period: Dose Escalation: Extension Phase
Arm/Group | Dose Escalation Part: E7016 4 mg/kg/Day + Temozolomide 150 mg/m^2 | Dose Escalation Part: E7016 8 mg/kg/Day + Temozolomide 150 mg/m^2
Started | 5 | 3
Completed | 3 | 2
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAS) consisted of all participants who received at least one dose of E7016 or temozolomide and had at least one safety assessment after receiving these medications.
Groups:
- Dose Escalation Part: E7016 4 mg/kg/Day + Temozolomide 150 mg/m^2: Participants received single oral dose of 4 mg/kg/day E7016 capsule on Day -7 for PK analysis, followed by once daily dose from days 1 to 5 in combination with temozolomide 150 mg/m^2 capsule and alone on days 6 and 7 of Cycle 1 (cycle length=28 days) in Treatment Phase. Participants who completed the Treatment Phase entered the Extension Phase of Dose Escalation Part and continued the treatment in Extension Phase in same manner of Treatment Phase until unacceptable toxicity, disease progression, termination by the treating investigator, withdrawal of consent, termination of the program by the sponsor, or treatment delay >2 weeks for recovery of toxicity.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Part: E7016 4 mg/kg/Day + Temozolomide 150 mg/m^2 | Dose Escalation Part: E7016 8 mg/kg/Day + Temozolomide 150 mg/m^2 | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (8.17) | 57.0 (8.19) | 55.3 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 8
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 7 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 2 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) for E7016 in Combination With Temozolomide
Description: The MTD was defined as the highest dose of E7016 in combination with temozolomide at which no more than one of six participants experienced a dose-limiting toxicity (DLT). DLTs were defined as those adverse events (AEs) considered related to E7016 which occurred during the first cycle of study drug administration. DLTs were evaluated and graded based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE version [v] 4.0).
Time Frame: Cycle 1 (Cycle length = 28 days)
Population: The SAS consisted of all participants who received at least one dose of E7016 or temozolomide and had at least one safety assessment after receiving these medications.
Measure: Number; unit: mg/kg/day
Groups:
- Dose Escalation Part, All Participants: E7016 + Temozolomide: Participants received single oral dose of 4 or 8 mg/kg/day E7016 capsule on Day -7 for PK analysis, followed by once daily dose from days 1 to 5 in combination with temozolomide 150 mg/m^2 capsule and alone on days 6 and 7 of Cycle 1 (cycle length=28 days) in Treatment Phase.
Arm/Group | Dose Escalation Part, All Participants: E7016 + Temozolomide
Number analyzed (Participants) | 12
mg/kg/day | 4

2. Primary Outcome: Number of Participants With Dose-limiting Toxicity (DLT)
Description: A DLT was defined as those AEs considered related to E7016 which occurred during the first cycle of study drug administration. DLTs were evaluated and graded based on the NCI CTCAE version 4.0. The following toxicities were regarded as DLTs: a Grade 4 hematologic toxicity (lasting [greater than or equal to] >=5 days); a temozolomide dose reduction for Grade >=3 neutropenia or thrombocytopenia; or a Grade >=3 nonhematologic toxicity (except optimally managed nausea, vomiting, or diarrhea) that was assessed by the investigator as related to study drug. A participant with two or more DLTs with the same preferred term was counted only once for that preferred term.
Time Frame: Cycle 1 (Cycle length = 28 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: E7016 4 mg/kg/Day + Temozolomide 150 mg/m^2 | Dose Escalation Part: E7016 8 mg/kg/Day + Temozolomide 150 mg/m^2
Number analyzed (Participants) | 9 | 3
Participants
  Tachycardia | 0 | 2
  Presyncope | 0 | 2
  Hypotension | 0 | 1

3. Primary Outcome: Alternative Dose of Interest (ADI) for E7016 in Combination With Temozolomide
Description: The ADI determination plan was based primarily on clinical, and/or PK measurements of drug concentration and/or bioactivity as defined by preclinical studies. However, the ADI was not pursued due to the limited sample size.
Time Frame: Cycle 1 (Cycle length = 28 days)
Population: An ADI was not pursued due to the limited sample size. No data was collected and analyzed to report in this outcome measure.
Arm/Group | Dose Escalation Part: E7016 4 mg/kg/Day + Temozolomide 150 mg/m^2 | Dose Escalation Part: E7016 8 mg/kg/Day + Temozolomide 150 mg/m^2
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR was defined as the percentage of participants with complete response (CR) plus partial response (PR) as determined by the investigator, using modified Response Evaluation Criteria in Solid Tumors (RECIST 1.1) in the evaluation of magnetic resonance imaging/computerized tomography (MRI/CT) scans of targeted lesions and photographs and bone scans if appropriate for the tumor type. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to less than 10 mm. PR was defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions. ORR = CR + PR
Time Frame: From Cycle 1 Day 1 up to 6 Cycles (Cycle length=28 days) of treatment, an average of 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Dose Escalation Part: E7016 4 mg/kg/Day + Temozolomide 150 mg/m^2 | Dose Escalation Part: E7016 8 mg/kg/Day + Temozolomide 150 mg/m^2
Number analyzed (Participants) | 9 | 3
Percentage of participants | 0.0 | 0.0

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who had BOR of CR plus PR plus stable disease (SD). The best observed response (BOR) was defined as the best response recorded from the start of the study treatment until discontinuation from the study. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions. SD was defined as nonCR/non-progressive disease (PD) (NN), for participants with nontarget lesions. The minimum duration of SD was 7 weeks of multiple dose treatment. For participants who did not have target lesions, the response category NN was used instead of SD. DCR = CR + PR + SD greater than or equal to 7 weeks
Time Frame: From Cycle 1 Day 1 up to 6 Cycles (Cycle length=28 days) of treatment, an average of 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Dose Escalation Part: E7016 4 mg/kg/Day + Temozolomide 150 mg/m^2 | Dose Escalation Part: E7016 8 mg/kg/Day + Temozolomide 150 mg/m^2
Number analyzed (Participants) | 9 | 3
Percentage of participants | 11.1 | 66.7

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the first dose of E7016 until 6 Cycles of treatment or death whichever occurs first.
Time Frame: From Cycle 1 Day 1 up to 6 Cycles (Cycle length=28 days) of treatment, an average of 24 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dose Escalation Part: E7016 4 mg/kg/Day + Temozolomide 150 mg/m^2 | Dose Escalation Part: E7016 8 mg/kg/Day + Temozolomide 150 mg/m^2
Number analyzed (Participants) | 9 | 3
days | 76.0 [16.0 to 267.0] | NA [121.0 to NA] — Median and upper limit of 95% Confidence Interval could not be determined due to insufficient number of deaths.

ADVERSE EVENTS:
Time Frame: From date of first dose up to 30 days after the last dose of study drug (up to 45 weeks)
Description: The SAS consisted of all participants who received at least one dose of E7016 or temozolomide and had at least one safety assessment after receiving these medications. As planned, combined safety data for Treatment phase and Extension phase was reported.
Arm/Group | Dose Escalation Part: E7016 4 mg/kg/Day + Temozolomide 150 mg/m^2 | Dose Escalation Part: E7016 8 mg/kg/Day + Temozolomide 150 mg/m^2
All-Cause Mortality (participants affected / at risk) | 4/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 5/9 | 1/3
Other Adverse Events (participants affected / at risk) | 9/9 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Part: E7016 4 mg/kg/Day + Temozolomide 150 mg/m^2 (N=9) | Dose Escalation Part: E7016 8 mg/kg/Day + Temozolomide 150 mg/m^2 (N=3)
Ascites (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 1
Disease progression (General disorders) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Hypovolemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Part: E7016 4 mg/kg/Day + Temozolomide 150 mg/m^2 (N=9) | Dose Escalation Part: E7016 8 mg/kg/Day + Temozolomide 150 mg/m^2 (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Palpitations (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 3
Periorbital oedema (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Addominal tenderness (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 3
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2
Asthenia (General disorders) | 2 | 0
Chest discomfort (General disorders) | 1 | 0
Fatigue (General disorders) | 5 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Candidiasis (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urine output decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 2
Paraethesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 2
Restless leg syndrome (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Mental status change (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea external (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated due to sponsor's strategic decision, which is unrelated to safety, therefore no participants were enrolled in the Dose Expansion part. Hence, no data collection and analysis were done during Dose Expansion part of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other